CLINICAL TRIAL: NCT01856179
Title: Accumulation of n-3 Long-chain (LC)-PUFA by Supplementation of SDA-rich Echium Oil in Humans Depending on Age, Gender and Physiological Stage
Brief Title: Supplementation of Land-based Stearidonic Acid (SDA)-Rich Oils in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil., University of Jena
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H42-KK
Record Dates: First submitted 2011-11-29; First posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Hypercholesterolemia; Overweight
Keywords: Conversion of ALA and SDA; Metabolism of n-3 fatty acids
MeSH Terms: conditions — Hypercholesterolemia; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Echium oil young (Experimental): BMI<25,
  age 20-30
  Interventions: Dietary Supplement: Echium oil
- Echium oil older (Experimental): age 40-70 BMI <25
  Interventions: Dietary Supplement: Echium oil
- Echium oil older, overweight (Experimental): age 40-70 BMI >25
  Interventions: Dietary Supplement: Echium oil

INTERVENTIONS:
Dietary Supplement: Echium oil — Oil of Echium platagineum (natural plant oil) ca. 15-18 g/d (Croda)

SUMMARY:
The objective of this study is to investigate the conversion of the precursors ALA and SDA into n-3 LC-PUFA (EPA, DPA and DHA) in humans by oral supplementation of Echium oil in comparison with SDA soybean oil (positive control). In addition, the accumulation of n-3 LC-PUFA is compared between subpopulations of different age, gender and physiological conditions (overweight, increased serum total cholesterol).

DETAILED DESCRIPTION:
N-3 PUFA are important for human health and nutrition. Due to the increasing world population, overfishing of the seas and generally low amounts of n-3 PUFA in major oil crops, there is a demand for new sources of n-3 PUFA.

One approach involves searching for potential vegetable sources of n-3 PUFA; especially those rich in ALA and SDA. The conversion of ALA to SDA in humans depends on the rate-limiting ∆6-desaturation. Plant-derived SDA is therefore a promising precursor regarding endogenous synthesis of n-3 LC-PUFA in humans. The enrichment of n-3 LC-PUFA in human lipids during the supplementation of ALA- and SDA-rich Echium oil will be compared with SDA-rich soybean oil.

Eighty volunteers will be recruited and allocated into four study groups depending on age and BMI. Three groups (each n=20) will receive daily ca. 20 g Echium oil ( group 1 and 2: mean BMI < 25, with mean age: 25 or 55 years; group 3: mean age 55 and BMI > 25). One group (n=20) will receive SDA soybean oil ( dose with comparable amount of SDA; BMI < 25; mean age 25 and 55). The double-blind, randomized, parallel-designed study will start with a two-weeks run-in period, followed by an eight-weeks supplementation period. After the run-in period, one week and eight weeks of oil supplementation blood will be drawn and 24-h urine will be sampled.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects

Exclusion Criteria:

* cholesterol lowering drugs
* chronic diseases
* pregnancy, lactation
* intake of nutritional supplements

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
eicosapentaenic acid | after 0,7, 56 days
  eicosapentaenic acid in lipids of plasma, erythrocytes and peripheral mononuclear cells (% of total identified fatty acid methyl esters)

SECONDARY OUTCOMES:
Lipid mediators derived from AA, EPA and DGLA such as HETE species (5-HETE; 8-HETE, etc.) | 0 and 56 days
  concentration in plasma (pg/µl plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Katrin Kuhnt, Dr. rer. nat, Principal Investigator — University of Jena, Insitute of Nutrition
Locations (1):
- Friedrich Schiller University of Jena, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Kuhnt K, Weiss S, Kiehntopf M, Jahreis G. Consumption of echium oil increases EPA and DPA in blood fractions more efficiently compared to linseed oil in humans. Lipids Health Dis. 2016 Feb 18;15:32. doi: 10.1186/s12944-016-0199-2. PMID 26892399
- [Derived] Kuhnt K, Fuhrmann C, Kohler M, Kiehntopf M, Jahreis G. Dietary echium oil increases long-chain n-3 PUFAs, including docosapentaenoic acid, in blood fractions and alters biochemical markers for cardiovascular disease independently of age, sex, and metabolic syndrome. J Nutr. 2014 Apr;144(4):447-60. doi: 10.3945/jn.113.180802. Epub 2014 Feb 19. PMID 24553695